CLINICAL TRIAL: NCT00947089
Title: The Role of Oxidized Regenerated Cellulose in Preventing Infections at the Surgical Site: Prospective, Randomized Study in 98 Patients Affected by a Dirty Wound
Brief Title: Role of Oxidized Regenerated Cellulose (ORC) Applied to "Dirty" Surgical Wounds
Acronym: ORC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Sergio Alfieri, UCSC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCSC 1
Record Dates: First submitted 2009-07-20; First posted 2009-07-27 (Estimated); Last update posted 2009-07-27 (Estimated); Status verified 2009-07

CONDITIONS: Infections
Keywords: ORC (oxidized regenerated cellulose); SSI (Surgical site infections)
MeSH Terms: conditions — Infections; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A-the treatment group (Experimental): Group A-patients have their wound, the site of the previous stoma, wad with ORC
  Interventions: Device: oxidized regenerated cellulose (Fibrillar SURGICEL)
- group B-the control group (Active Comparator): control group-patients have their wound wad with iodoform gauze
  Interventions: Device: iodoform gauze

INTERVENTIONS:
Device: oxidized regenerated cellulose (Fibrillar SURGICEL) — one gauze made of ORC
  Other Names: Fibrillar SURGICEL (Ethicon, Somerville, New Jersey)
  Arms: group A-the treatment group
Device: iodoform gauze — one iodoform gauze
  Arms: group B-the control group

SUMMARY:
The purpose of this study is to determine whether oxidized regenerated cellulose (ORC) is effective to reduce the risk of surgical site infections (SSI).

DETAILED DESCRIPTION:
Surgical site infections (SSI) have significant clinical and economic repercussions since they still are the most common cause of nosocomial infections in surgical patients. It is important to bear in mind the growing number of SSI due to antibiotic-resistant microorganisms.

ELIGIBILITY:
Inclusion Criteria:

* have an ileostomy or a colostomy
* are candidates for an elective surgical procedure of ostomy closure

Exclusion Criteria:

* immunodeficiency
* chronic use of corticosteroids or antibiotics
* chemotherapy and/or radiotherapy in the last 30 days before closure of the stoma
* concomitant foci of infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2003-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
to reduce the microbial load and, consequently, the infection rate as compared to conventional local wound treatment | third post-operative day

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Alfieri, MD, Study Chair — UCSC
Locations (1):
- Digestive Surgery of the Catholic University of Sacred Heart, Rome, Italy